CLINICAL TRIAL: NCT03280641
Title: The Role of D-dimer in Patients With Atrial Fibrillation Receiving Anticoagulation Therapy
Brief Title: D-dimer In Patients With atRial Fibrillation rEceiving antiCoagulation Therapy
Acronym: DIRECT
Status: Completed | Type: Observational
Sponsor: Wuhan Asia Heart Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-P-016
Record Dates: First submitted 2017-09-10; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Atrial Fibrillation; Strokes Thrombotic
MeSH Terms: conditions — Atrial Fibrillation; Thrombotic Stroke | interventions — Dabigatran; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dabigatran Group: Patiets with atrial fibrillation received dabigatran (110mg, bid).
  Interventions: Drug: Dabigatran Etexilate 110mg
- Warfarin Group: Patiets with atrial fibrillation received warfarin (110mg, bid).The target international normalized ratio (INR):1.6-3.0
  Interventions: Drug: Warfarin Sodium

INTERVENTIONS:
Drug: Dabigatran Etexilate 110mg — Dabigatran Etexilate 110mg, BID
  Other Names: Pradaxa
  Groups: Dabigatran Group
Drug: Warfarin Sodium — Target INR:1.6-3.0
  Groups: Warfarin Group

SUMMARY:
This is a sigle-center, prospective study to evaluate the role of D-Dimer testing in patients with atrial fibrillation receiving Dabigatran or warfarin anticoagulation therapy.

DETAILED DESCRIPTION:
Patients with atrial fibrillation receiving Dabigatran or warfarin anticoagulation therapy was screened and signed to two group: Dabigatran group and Warfarin group. D-dimer test was analyzed before and 3 months after anticoagulation starting specificly. Patients were followed-up for at least 12 months,and clinical outcomes, including thrombotic events major bleeding events and all-cause deaths were recorded during follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Non-valvular atrial fibrillation
* Receiving oral anticoagulation therapy and have good compliance

Exclusion Criteria:

* Life expectancy less than 1 year
* Thrombosis or major bleeding history within 3 months
* Refusal to Participate

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Non-valvular atrial fibrillation receiving Dabigatran or warfarin anticoagulation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 1194 (Actual)
Dates: Start 2015-08-09 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Cardiovascular events | 12 months
  Thrombotic events, cardiovascular deaths, major bleeding events

CONTACTS AND LOCATIONS:
Overall Officials: Litao ZHANG, MD, Principal Investigator — Wuhan Asia Heart Hospital
Locations (1):
- WAHH, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
We will share the IPD after the paper being published